CLINICAL TRIAL: NCT01561404
Title: Effect of the Inhibition of the Mammalian Target of Rapamycin on Metabolism and Exercise.
Acronym: EXETOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of potential patients
Sponsor: Josep M Cruzado (Other)
Responsible Party: Sponsor-Investigator, Josep M Cruzado, NEPHROLOGIST, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MTOR-METAB; 2009-010541-31 (EudraCT Number)
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Disorder Related to Renal Transplantation; Exercise, Aerobic; Muscle Strength
MeSH Terms: conditions — Motor Activity | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): Conversion from calcineurin inhibitor (CNI) to MTOR inhibitor (everolimus)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — In patients that change of immunosuppressive therapy from calcineurin inhibitor (CNI)(tacrolimus or cyclosporine) to m-TOR (everolimus)has been clinically indicated, check if there is an increase in physical exercise capacity.
  Other Names: m-TOR inhibitor(Everolimus)in kidney transplant recipients

SUMMARY:
This is an exploratory study based on the hypothesis that kidney transplant patients treated with an immunosuppressive therapy based on an inhibitor of the mammalian target of rapamycin (m-TOR) may increase resistance to physical exercise, which would result in an improvement in the quality of life of these patients.

DETAILED DESCRIPTION:
The hypothesis of the present study is that, with respect to calcineurin inhibitors, the mTOR inhibitor-based immunosuppression may alter the physical exercise capacity in renal transplant patients.

This is based on recent data obtained. Regarding metabolism there is evidence that inhibition of mTOR, reduces muscle glucose utilization, as well as, increase fatty acid oxidation. On the other hand, has shown that drugs based on mTOR inhibitors in the context of excess of nutrients improves intracellular glucose uptake in skeletal muscle cells. Through these mechanisms could increase resistance to physical exercise, which would result in an improvement in the quality of life of patients. Nevertheless, there isn't any paper that has explored this hypothesis accurately.

ELIGIBILITY:
Inclusion Criteria:

1. Renal transplant patient's aged between 18 and 60 years old.
2. Heart rate in radial pulse and seated between 50 and 100 bpm.
3. Systolic blood pressure between 100 and 140 and diastolic between 50 to 90.
4. Absence of any clinical physical, psychological or psychiatric condition that would prevent from the protocol described follow-up.
5. Estimated glomerular filtration rate greater than 40 ml / min.
6. Proteinuria < 0.5 g / d.
7. Renal transplantation at least 6 months ago.
8. Immunosuppressant based on calcineurin inhibitors.
9. Hemoglobin > 11 g / dl.
10. Body mass index (BMI) < 35 kg/m2.
11. Indication for conversion to everolimus and granting of written informed consent.

Exclusion Criteria:

1. Diabetes mellitus
2. Treatment with erythropoiesis stimulating drugs
3. Treatment with β blockers drugs
4. Participation in any clinical trial in the last 30 days prior to the inclusion.
5. Any other physical illness, psychological or psychiatric condition that could difficult the follow-up of the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Muscular strength | Change from baseline to 6-8 weeks after m-TOR conversion
  The principal variable is the increase of the exercise capacity measured by 2 sub-varibles: muscular strenght and decrease of oxygen consumption in the tissues.
Oxygen consumption in the tissues | Change from baseline to 6-8 weeks after m-TOR conversion
  The principal variable is the increase of the exercise capacity measured by 2 sub-varibles: muscular strenght and decrease of oxygen consumption in the tissues.

SECONDARY OUTCOMES:
Anthropometric measures | Change from baseline to 6-8 weeks after m-TOR conversion
  Measure of anthropometric measures including height,weight, muscular folds( biceps, triceps, subscapular, pectoral, axillary, abdominal, suprailiac, thigh and leg) and perimeters (arm, forearm, wrist, abdominal, waist, hip, thigh, groin, thigh and leg).
Strength of the hand | Change from baseline to 6-8 weeks after m-TOR conversion
  Measure of the strenght of the hand will include:test of maximum strength of contraction of the palm, maximum resistance force of the palm and maximum power on a cycle ergometer for 5 seconds with a constant resistance of 50 N.
Metabolic parameters- Cardioventilatory response | Change from baseline to 6-8 weeks after m-TOR conversion
  Cardioventilatory response measured with respiratory rate, ventilation, oxygen consumption, carbon dioxide production, respiratory quotient and tidal volume during stress test.
Metabolic parameters- Biochemical response | Change from baseline to 6-8 weeks after m-TOR conversion
  Lactate and blood glucose levels after stress test
Glucose tolerance test | Change from baseline to 6-8 weeks after m-TOR conversion
Blood pressure | Change from baseline to 6-8 weeks after m-TOR conversion
  Continuos blood preassure measure (24 hours) with a holter monitor device.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M. Cruzado, MD, Principal Investigator — Nephrology Department Hospital Universitari de Bellvitge
Locations (1):
- Nephrology Department. Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelone, Spain